CLINICAL TRIAL: NCT00976495
Title: An Exploratory Phase 2 Study to Assess the Effect of Dapagliflozin on Glomerular Filtration Rate (GFR) in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic and Blood Pressure (BP) Control
Brief Title: Effects of Dapagliflozin on Kidney Function (Glomerular Filtration Rate) in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Astra Zeneca, Bristol-Myers Squibb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MB102-035; EUDRACT #: 2009-010221-39
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Placebo
- Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, once daily, 12 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 12 weeks
  Arms: Dapagliflozin
Drug: Hydrochlorothiazide — Tablets, Oral, 25 mg, once daily, 12 weeks
  Arms: Hydrochlorothiazide

SUMMARY:
The purpose of this study is to evaluate the effects of dapagliflozin on kidney function, as assessed by glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes and inadequate glycemic control, defined as A1C ≥ 6.6 and ≤ 9.5%
* Stable dose of metformin AND/OR a sulfonylurea, for at least 4 weeks prior to the enrollment visit
* Inadequate blood pressure (BP) control, defined as systolic BP (SBP) ≥ 130 and < 165 mmHg, AND/OR diastolic BP (DBP) ≥ 80 and < 105 mmHg
* C-peptide ≥ 0.8 ng/mL
* Estimated GFR by the Modification of Diet in Renal Disease (MDRD) formula > 60 mL/min/1.73m² and < 150 mL/min/1.73m²
* Urine albumin:creatinine ratio (UACR) < 300 mg/g
* BMI ≤ 45.0 kg/m2

Exclusion Criteria:

* Administration of diuretics or other medication approved for the treatment of hypertension (with the exception of either ACEI or ARB), at any dose during the 12 weeks prior to the enrollment visit
* History of adverse reaction to radio-contrast dye
* Allergy or contraindication to use of thiazide diuretics
* Aspartate Aminotransferase (AST) > 3X Upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 3X ULN
* Serum Total Bilirubin > 1.5X ULN
* Serum Creatinine (Scr) ≥ 1.50 mg/dL (133 μmol/l) for men; SCr ≥ 1.40 mg/dL (124 μmol/l) for women
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncologic, endocrine, psychiatric, or rheumatic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (9):
  - Advanced Clinical Res Inst, Anaheim, California
  - Torrance Clinical Research, Lomita, California
  - Elite Research Institute, Miami, Florida
  - Compass Research, Llc, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - University Of Michigan, Ann Arbor, Michigan
  - Prism Research, Saint Paul, Minnesota
  - Memorial Hospital Of Rhode Island, Pawtucket, Rhode Island
  - Zablocki Veterans Affairs Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - Local Institution, Toronto, Ontario
  - Local Institution, Laval, Quebec
- Local Institution, Groningen, Netherlands

REFERENCES:
- See also: Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3906841/
- See also: MB102035_Redacted_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3641&filename=MB102035_Redacted_CSR_synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 154 participants enrolled, 77 completed a qualification period. Of these 77 participants, 75 were randomized and received treatment. Of these 75 participants, 74 completed double-blind treatment period.
Groups:
- Placebo; Dapagliflozin 10 mg; Hydrochlorothiazide 25 mg: Tablet, oral, once daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Started | 25 | 24 | 26
Completed | 25 | 23 | 26
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg | Total
Number analyzed (Participants) | 25 | 24 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (9.50) | 53.7 (9.38) | 54.8 (9.87) | 55.5 (9.63)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 19 | 22 | 21 | 62
  65 - 75 years | 6 | 2 | 5 | 13
Sex/Gender, Customized [Number; unit: Participants]
  Male | 18 | 16 | 15 | 49
  Female | 7 | 8 | 11 | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 17 | 19 | 20 | 56
  Black/African American | 4 | 4 | 4 | 12
  Asian | 3 | 0 | 2 | 5
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Percent Change From Baseline in Glomerular Filtration Rate (GFR) at Week 12 (Modified Last Observation Carried Forward [MLOCF])
Description: Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. If no Week 12 measurement was available, the last available post-baseline measurement obtained on or after Day 23 was used regardless of rescue medication. Measurements were obtained during radomization visit, and Week 12 in the double-blind period by a central laboratory.
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 12 (MLOCF)
Measure: Mean (Standard Error); unit: % Change of Baseline GFR
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Number analyzed (Participants) | 25 | 22 | 26
% Change of Baseline GFR | -2.92 (2.0133) | -10.76 (1.9684) | -3.40 (1.9756)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -8.07, 95% CI 2-sided [-13.34 to -2.49], Standard Error of Mean 2.7177 — ANCOVA was applied. Given that this was a pilot study designed for exploratory analysis, formal statistical hypothesis testing was not performed
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Hydrochlorothiazide 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -7.62, 95% CI 2-sided [-12.87 to -2.06], Standard Error of Mean 2.7068 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Adjusted Mean Change From Baseline in 24-Hour Ambulatory Systolic Blood Pressure (ASBP) at Week 12 (Last Observation Carried Forward [LOCF])
Description: Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Measurements were obtained during lead-in, and Week 12 in the double-blind period.
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing ASBP values at baseline and Week 12 (LOCF)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Number analyzed (Participants) | 25 | 22 | 25
mmHg | -0.88 (1.6373) | -3.28 (1.7674) | -6.55 (1.6833)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.40, 95% CI 2-sided [-7.11 to 2.31], Standard Error of Mean 2.3613 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Hydrochlorothiazide 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.26, 95% CI 2-sided [-1.55 to 8.08], Standard Error of Mean 2.4112 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Adjusted Mean Change From Baseline in Daytime (0900 to 2100 Hours) Ambulatory Systolic Blood Pressure (ASBP) at Week 12 (Last Observation Carried Forward [LOCF])
Description: as for outcome 2
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing ASBP values at baseline and Week 12 (LOCF)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Number analyzed (Participants) | 25 | 22 | 25
mmHg | -1.55 (1.7247) | -5.93 (1.8673) | -6.83 (1.7671)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-9.38 to 0.63], Standard Error of Mean 2.5072 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Hydrochlorothiazide 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-4.18 to 5.99], Standard Error of Mean 2.5474 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Adjusted Mean Change From Baseline in Nighttime (0100 to 0600 Hours) Ambulatory Systolic Blood Pressure (ASBP) at Week 12 (Last Observation Carried Forward [LOCF])
Description: as for outcome 2
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing ASBP values at baseline and Week 12 (LOCF)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Number analyzed (Participants) | 25 | 22 | 25
mmHg | -0.61 (1.9468) | -0.45 (2.0822) | -7.76 (1.9857)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-5.39 to 5.71], Standard Error of Mean 2.7812 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Hydrochlorothiazide 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.31, 95% CI 2-sided [1.70 to 12.93], Standard Error of Mean 2.8135 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 12 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo | Dapagliflozin 10 mg | Hydrochlorothiazide 25 mg
Serious Adverse Events (participants affected / at risk) | 0/25 | 3/24 | 0/26
Other Adverse Events (participants affected / at risk) | 2/25 | 6/24 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dapagliflozin 10 mg (N=24) | Hydrochlorothiazide 25 mg (N=26)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dapagliflozin 10 mg (N=24) | Hydrochlorothiazide 25 mg (N=26)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2) | 4 (4)
MALAISE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No